CLINICAL TRIAL: NCT03831776
Title: A Study of Efficacy and Safety of Long-acting Low Dose Ropeginterferon in Patients With Chronic Myeloid Leukemia Treated With Bosutinib From Diagnosis: a Randomized Prospective Trial
Brief Title: Long-acting Low Dose Ropeginterferon for Chronic Myeloid Leukemia Treated With Bosutinib From Diagnosis
Acronym: BosuPeg
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: St. Olavs Hospital (Other)
Collaborators: Haukeland University Hospital (Other); Oslo University Hospital (Other); University Hospital of North Norway (Other); Helse Stavanger HF (Other Government); Henri Mondor University Hospital (Other); Hôpital René Huguenin (Unknown); Hôpital Mignot, Versailles Paris (Unknown); Uppsala University Hospital (Other); Odense University Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: BosuPeg TRIAL; 2018-001044-54 (EudraCT Number)
Record Dates: First submitted 2019-02-04; First posted 2019-02-06 (Actual); Last update posted 2025-06-08 (Actual); Status verified 2025-06

CONDITIONS: Chronic Myeloid Leukemia
Keywords: Bosupeg; Ropeginterferon
MeSH Terms: conditions — Leukemia, Myelogenous, Chronic, BCR-ABL Positive | interventions — bosutinib

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Bosutinib-Ropeginterferon combination (Experimental)
  Interventions: Drug: Bosutinib; Drug: Ropeginterferon
- Bosutinib monotherapy (Active Comparator)
  Interventions: Drug: Bosutinib

INTERVENTIONS:
Drug: Bosutinib — Bosutinib, provided by Pfizer, starting dose of 200mg QD and stepwise dose escalation (> 300 mg/d > 400 mg/d) during the first three months. A pharmacological study will be performed in the French cohort (BOSUSTEP Substudy). BOS residual plasma concentration (Cmin) will be checked after initiation, before each dose step in the French cohort, and at M3 also for Nordic patients in ancillary studies.
Drug: Ropeginterferon — Ro-Peg-Interferon α2b will be supplied by AOP Orphan to be administered by subcutaneous injections from prefilled injection pens. RoPegIFN will be given in an open-label fashion. Patients assigned to RoPegIFN will start with 50 μg injected subcutaneously every 14 days, in combination with Bosutinib.
  Other Names: RoPegIFN
  Arms: Bosutinib-Ropeginterferon combination

SUMMARY:
To study the efficacy and safety of combination of Ro-Peg-interferon-α2b (RoPegIFN) with Bosutinib (BOS) in comparison to BOS monotherapy, as frontline therapy for newly diagnosed chronic myeloid leukemia patients, and to estimate efficacy of the addition of RoPegIFN to BOS in terms of deep molecular response with the aim of increasing the proportion of patients who may achieve treatment free remission. (NCMLSG study #NordCML012)

ELIGIBILITY:
Inclusion Criteria:

* Signed written informed consent form (ICF) before any procedure related to the study
* Newly diagnosed (≤ 3 months) BCR-ABL positive chronic myeloid leukemia (CML) in chronic phase
* Major BCR-ABL transcripts (p210 b2a2(e13a2) and/or b3a2 (e14a2)
* Not previously treated for CML except with hydroxyurea or anagrelide
* ECOG Performance Status (ECOG PS) ≤ 2
* Adequate organ function: Total bilirubin < 1,5 times the institutional Upper Limit of Normal (ULN); Hepatic enzymes ASAT and ALAT < 2 times the institutional ULN; Serum Creatinine < 1.5 time the institutional ULN; Lipase < 1.5 time the institutional ULN
* Women of childbearing potential (WOCBP) must be using an adequate method of contraception to avoid pregnancy throughout the study.
* WOCBP must have a negative serum or urine pregnancy test at screening.
* Free subject, without guardianship nor subordination
* Health insurance coverage

Exclusion Criteria:

* Patients with BCR-ABL transcript other than M-BCR-ABL
* Patients previously treated with tyrosine kinase inhibitors (TKIs).
* Inability to freely provide consent through judiciary or administrative condition.
* Ongoing participation to another clinical investigational study.
* Medical history and concurrent diseases: a) Hypersensitivity to any of the excipients of BOS or RoPegIFN, b) Prior treatment with Interferon-α, contraindication to interferon-α, c) Autoimmune disorder, concomitant immunosuppressive treatment or corticosteroids, d) Pre-existing thyroid disease unless controlled with conventional treatment, auto-immune thyroiditis, e) Chronic liver disease, f) Prior or ongoing severe psychiatric disease, g) HIV positivity, chronic hepatitis B or C, h) Uncontrolled or severe cardiac (NYHA Class III or IV) or pulmonary disease, echocardiography with LVF < 45% or LLN, peak velocity of tricuspid regurgitant flow > 2,8 m/s, pulmonary arterial hypertension (PAH), QTc>450 ms (by Barrets correction)
* Other malignant disease during the last 5 years prior to the inclusion except non-melanoma skin carcinoma or carcinoma in situ of the cervix,
* History of significant bleeding disorder unrelated to CML or diagnosed congenital bleeding disorder,
* Subjects with an uncontrolled undercurrent illness or any concurrent condition that, in the investigator's opinion, would jeopardize the safety of the subject or compliance with the protocol.
* Prohibited treatments and/or therapies: strong inhibitors/inducers of the CYP 3A4,
* History / any condition for poor compliance to medical treatment.
* Women who are pregnant or breastfeeding are not eligible for this study

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 212 (Actual)
Dates: Start 2019-03-25 (Actual); Primary Completion 2024-12-31 (Actual); Study Completion 2024-12-31 (Actual)

PRIMARY OUTCOMES:
Rate of molecular response 4 (MR4) | 12 months
  Molecular response 4 (MR4) is defined by either a positive BCR-ABL/ABL ratio ≤ 0.01% on the international scale (IS) or by undetectable BCR-ABL with the analysis of at least 10000 copies of ABL or 24000 copies of GUS (according to the ELN recommendations by N. Cross et al., Leukemia 2015)

SECONDARY OUTCOMES:
Rate of molecular response MR2, MR3, MR4, MR4.5 from 1 month up to 24 months and every 6 months thereafter | 2 years
Cumulative incidence of molecular response MR3, MR4, MR4.5 | 2 years
Rate of complete cytogenetic response (CCyR) up to 12 months | 12 months
Rate of undetectable molecular response for patients who achieved molecular response MR4 and MR4.5 | 2 years
Time to and duration of CCyR, MR3, MR4, MR4.5 | 2 years
proportion of patients eligible for randomization after 3 months of Bosutinib | 3 months
rate and characteristics of severe adverse events (SAE) | 2 years
  type and grade according to the NCI CTCAE v4.03
Dose intensity of RoPegIFN and Bosutinib | 2 years
Cumulative incidence of discontinuation of the therapies, incl. reasons for discontinuation | 2 years
Quality of life assessment by QLQC30 questionnaire up to 6 years at key time point (Day 1, month 3, month 6, month 12, month 24, month 48, month 54, month 72) | 6 years
Quality of life assessment by CML24 questionnaire up to 6 years at key time point (Day 1, month 3, month 6, month 12, month 24, month 48, month 54, month 72) | 6 years
The proportion of patients achieving a durable deep molecular response and being eligible for treatment discontinuation at month 48 | 4 years
  Sustained deep molecular response (MR) criteria will be defined according updated data and ELN guidelines before the first patient will achieve month 48 (at least a MR4 over a 12 months period and confirmed on the last centralized measurement at month 48

CONTACTS AND LOCATIONS:
Overall Officials: Tom Christian Martinsen, md phd, Study Director — St Olavs Hospital, Clinical of Internal Medicine; Henrik Hjorth-Hansen, md phd, Principal Investigator — St. Olavs Hospital; Lydia Roy, md phd, Principal Investigator — Centre Hospitalo-Universitaire Henri Mondor, Service d'Hematologie Clinique
Locations (18):
- Denmark (4):
  - Aalborg university hospital, Aalborg
  - Aarhus ..., Aarhus
  - Copenhagen ..., Copenhagen
  - Odense Universitetshospital, Odense
- Comprehensive Cancer Center, Hematology, Helsinki, Finland
- Norway (5):
  - Haukeland Universitetssjukehus, Bergen
  - Oslo Universitetssykehus, Oslo
  - Stavanger Universitetssjukehus, Stavanger
  - Universitetssykehuset Nord Norge, Tromsø
  - St Olavs Hospital, Trondheim
- Sweden (8):
  - Göteborg ...., Gothenburg
  - Universitetssjukhuset Linköping, Linköping
  - Skåne University Hospital, Lund
  - Universitetssjukhuset Örebro, Örebro
  - Karolinska Universitetssjukhus, Stockholm
  - Sundsvall ..., Sundsvall
  - Norrlands Universitetssjukhus, Umeå
  - University Hospital, Uppsala